CLINICAL TRIAL: NCT01968382
Title: A Multicenter Randomized, Double-Blind, Placebo-controlled, Dosing, Safety and Efficacy Study of IMM 124-E (Hyperimmune Bovine Colostrum) for Patients With Severe Alcoholic Hepatitis
Brief Title: Safety and Efficacy of IMM 124-E for Patients With Severe Alcoholic Hepatitis
Acronym: TREAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Immuron Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20000157; U01AA021891 (NIH); IMM-124-E (Other: VCU)
Record Dates: First submitted 2013-08-30; First posted 2013-10-24 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis, Alcoholic
Keywords: IMM 124-E; Bovine Colostrum; Alcoholic; Hepatitis; LPS; Hyper-immune
MeSH Terms: conditions — Hepatitis, Alcoholic; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IMM 124-E 2400 mg/day (Experimental): Imm-124-E (2400 mg/day) will be provided in two divided doses daily in the form of powder to be mixed with water. Subjects will get 1 active drug powder and 1 placebo powder with each dosing for a total of 4 sachets daily.
  Interventions: Drug: IMM 124-E (Hyperimmune Bovine Colostrum); Drug: Placebo (High protein milk powder)
- IMM 124-E 4800 mg/day (Experimental): Imm-124-E (4800 mg/day) will be provided in two divided doses daily in the form of 2400 mg in the form of a powder to be mixed with water. The total number daily will be 4 sachets.
  Interventions: Drug: IMM 124-E (Hyperimmune Bovine Colostrum)
- Placebo (High protein milk powder) (Placebo Comparator): Subjects will receive 2 sachets of placebo powder to be mixed with water in the morning and 2 sachets of placebo powder (to be mixed with water) in the evening for a total of 4 sachets of placebo daily.
  Interventions: Drug: Placebo (High protein milk powder)

INTERVENTIONS:
Drug: IMM 124-E (Hyperimmune Bovine Colostrum) — Hyper-immune bovine colostrum enriched with anti-LPS antibodies and which has been designated by Immuron as IMM-124E.
  Arms: IMM 124-E 2400 mg/day; IMM 124-E 4800 mg/day
Drug: Placebo (High protein milk powder) — Subjects will receive a total of 4 sachets (2 in the morning and 2 in the evening) daily
  Arms: IMM 124-E 2400 mg/day; Placebo (High protein milk powder)

SUMMARY:
Hypothesis: Oral administration of hyperimmune bovine colostrum enriched with anti-LPS antibodies will reduce endotoxemia, and improve pathophysiological and clinical parameters related to severe alcoholic hepatitis (SAH).

IMM 124-E is safe in subjects with severe alcoholic hepatitis being treated with steroids.

Aim: To perform a phase 2a "proof of concept" placebo-controlled, dose-ranging study of Imm 124-E (hyperimmune bovine colostrum enriched with IgG anti-LPS) in subjects with severe AH on steroids.

DETAILED DESCRIPTION:
Subjects with severe alcoholic hepatitis (20=> MELD <=28) about to receive prednisolone (40 mg/day x 28 days) will be randomized 1:1:1 to additionally receive either one of two doses of IMM 124-E (2400 mg/day or 4800 mg/day) orally or placebo for the same duration. Standard of care nutrition support and alcohol cessation recommendations will be provided to all subjects. Alcohol withdrawal will be managed per standard of care. Subjects who meet Lille criteria for failure of treatment on day 7 or side effects requiring discontinuation of steroids will be removed from the study. The primary endpoint is a decrease in plasma endotoxin levels.

The secondary endpoints will include:

1. Mechanistic endpoints: TNF-α, immune-inflammatory markers, microbiome-metagenome
2. Efficacy-related: number of subjects meeting Lille failure criteria at day 7 , mortality (at 30 days, 90 days, and 180 days), time to drop in conjugated bilirubin by 50%, bile acids, liver function tests, change in MELD, and sequential organ failure
3. Safety related: tolerability, adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic hepatitis
* Men and women age 21 and above
* MELD >= 20 but <=28
* About to initiate prednisolone treatment, < 7 days of steroid treatment, or treatment naive.
* Actively consuming alcohol within 6 weeks of entry into the study
* Willing and able to comply with study requirements (including contraception)
* Subjects or their legally authorized representative (LAR) who have provided voluntary written informed consent.

Exclusion Criteria:

* Failure to obtain informed consent
* Subjects who are known to be HIV positive
* Active infection or sepsis (pneumonia by X-ray, positive blood or urine culture) or multi-organ failure
* Other or concomitant liver disease present: viral hepatitis, autoimmune liver disease, metabolic liver disease, vascular liver disease
* Cow milk allergy or severe lactose intolerance
* Active GI bleeding
* Untreated spontaneous bacterial peritonitis based on >250 polymorphonuclear cells or positive culture
* Acute kidney injury at time of randomization with Creatinine > 1.5 md/dL
* Evidence of acute pancreatitis (by imaging and lipase) or biliary obstruction (dilated bile ducts)
* Subjects who are pregnant or lactating
* Significant systemic or major illness, that, in the opinion of the Investigator would preclude the patient from participating in and completing the study
* Patients requiring the use of vasopressors or inotropic support in 12 hours prior to randomization
* Treatment for alcoholic hepatitis within 1 month of study entry with corticosteroids use>1 week immediately prior to the time of entry into the study.
* Any patient who has received any investigational drug or device within 30 days of dosing or who is scheduled to receive another investigational drug or device in the course of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-12; Primary Completion 2018-12-22 (Actual); Study Completion 2018-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun J Sanyal, MBBS MD, Principal Investigator — Virginia Commonwealth University
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Started | 18 | 19 | 20
Completed | 18 | 19 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder) | Total
Number analyzed (Participants) | 18 | 19 | 20 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (10.2) | 44.4 (11) | 45.7 (11.8) | 44.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 8 | 26
  Male | 10 | 9 | 12 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 13 | 18 | 17 | 48
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 20 | 57

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal Safety Endpoints
Description: Number of events and severity of gastrointestinal events, including nausea, vomiting, and diarrhea
Time Frame: 30 Days
Measure: Number; unit: Incidents
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 18 | 19 | 20
Incidents
  Mild | 15 | 27 | 7
  Moderate | 14 | 25 | 18
  Severe | 5 | 3 | 6

2. Primary Outcome: Combined Kidney, Brain, and Lung Safety Endpoints
Description: Number of incidents of the following: renal failure, encephalopathy or pulmonary compromise.
Time Frame: 30 Days
Measure: Number; unit: incidents
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 18 | 19 | 20
incidents
  Renal failure | 9 | 10 | 11
  Encephalopathy | 0 | 1 | 0
  Pulmonary compromise | 5 | 6 | 8

3. Primary Outcome: Infection Safety Endpoints
Description: Number of incidents of sepsis.
Time Frame: 30 Days
Measure: Number; unit: Incidents
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 18 | 19 | 20
Incidents | 2 | 1 | 2

4. Primary Outcome: Other Safety Endpoints
Description: Number of incidents of all other serious adverse events and other adverse events not already assessed as a primary outcome.
Time Frame: 30 Days
Measure: Number; unit: Events
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 18 | 19 | 20
Events | 67 | 113 | 124

5. Secondary Outcome: Bowel Gastrointestinal Safety Endpoints
Description: Number of participants who experience diarrhea
Time Frame: 30 Days
Population: Data were not collected separately for participants who suffered diarrhea. All gastrointestinal events (including diarrhea) were recorded as generic gastrointestinal events and reported in primary outcome #1.
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Circulating Endotoxin Levels
Description: Changes in endotoxin levels as measured using a standard blood assay
Time Frame: Baseline, day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 18 | 19 | 20
ng/mL | -361.06 (1249.17) | -72.94 (755.23) | 123.41 (469.38)
Statistical Analysis 1: Comparison: IMM 124-E 2400 mg/Day vs IMM 124-E 4800 mg/Day vs Placebo (High Protein Milk Powder); Test type: Superiority; p = 0.3198, ANOVA

7. Secondary Outcome: Lille Model Score
Description: Number of participants who meet Lille criteria indicating failure to respond to treatment
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 17 | 19 | 19
Participants | 5 | 6 | 9

8. Secondary Outcome: Mortality
Description: Number of deaths due to any cause
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 18 | 19 | 20
Participants | 5 | 2 | 2

9. Secondary Outcome: Change in Liver Function
Description: Model for end-stage liver disease (MELD) score ranges from 6 to 40 with higher number indicating worse liver function.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 9 | 11 | 9
score on a scale | -8.89 (5.35) | -6.82 (4.87) | -7.78 (12.12)
Statistical Analysis 1: Comparison: IMM 124-E 2400 mg/Day vs IMM 124-E 4800 mg/Day vs Placebo (High Protein Milk Powder); Test type: Superiority; p = 0.8462, ANOVA

10. Secondary Outcome: SOFA Score
Description: SOFA is a single score based on patient status of six different biological systems: respiratory, cardiovascular, hepatic, coagulation, renal, and neurological. Scores range from 0 to 24 with higher scores indicated worse status.
Time Frame: 30 days
Population: Data not collected
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change in Serum Bile Acids
Description: Serum bile acids levels as measured using standard blood serum assay
Time Frame: Baseline to 90 days
Population: Data not collected
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Time to 50% Drop in Bilirubin
Description: Length of time to a drop in bilirubin of 50% measured in days
Time Frame: 180 days
Population: Data not collected
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Cytokine Data
Description: Changes in cytokine profile across study arms at day 28
Time Frame: 28 days
Population: Data not collected
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment until 24 weeks following the initial dose of study medication.
Description: An adverse event is any untoward medical occurrence in a subject participating in a clinical trial. This includes any unfavorable and unintended sign, symptom or disease temporally associated with the use of the study medication, whether or not considered related to the study medication. This definition also includes accidental injuries, reasons for any change in medication, reasons for hospital admission, or reasons for surgical procedures.
Arm/Group | IMM 124-E 2400 mg/Day | IMM 124-E 4800 mg/Day | Placebo (High Protein Milk Powder)
All-Cause Mortality (participants affected / at risk) | 5/18 | 2/19 | 2/20
Serious Adverse Events (participants affected / at risk) | 11/18 | 9/19 | 12/20
Other Adverse Events (participants affected / at risk) | 18/18 | 19/19 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM 124-E 2400 mg/Day (N=18) | IMM 124-E 4800 mg/Day (N=19) | Placebo (High Protein Milk Powder) (N=20)
hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
perforated ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0)
hepatic encephalopathy (Nervous system disorders) | 3 (3) | 1 (1) | 3 (4)
sepsis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
alcohol withdrawal syndrome (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
blood creatinine abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
alcohol use (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
idiosyncratic alcohol intoxication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (2)
hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
renal injury (Renal and urinary disorders) | 1 (1) | 2 (3) | 1 (1)
hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
fluid imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
endotracheal intubation (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
multi-organ failure (General disorders) | 1 (1) | 2 (2) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (5)
blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ascites (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (2)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
explorative laparotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
liver transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
lobar pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM 124-E 2400 mg/Day (N=18) | IMM 124-E 4800 mg/Day (N=19) | Placebo (High Protein Milk Powder) (N=20)
urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Oedema (General disorders) | 2 (2) | 1 (1) | 2 (2)
renal injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 5 (5)
phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 2 (3)
laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
psychogenic seizure (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
transaminases increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
varices oesophageal (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
oral fungal infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 4 (4)
protein c deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
oedema peripheral (General disorders) | 4 (6) | 5 (9) | 5 (6)
central venous catheterisation (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
bladder catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
debridement (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
antiphospholipid antibodies positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
lesion excision (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — mixed respiratory and metabolic
mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
culture wound positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 3 (4)
bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
chills (General disorders) | 0 (0) | 3 (4) | 2 (2)
tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (2) | 5 (5) | 0 (0)
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
tongue abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 0 (0)
hyperammonaemia (Investigations) | 3 (3) | 0 (0) | 1 (2)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 3 (4) | 5 (7) | 0 (0)
hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
ascites (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2)
asterixis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3)
jaundice (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
insomnia (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0)
oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (4)
ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 2 (3)
glomerular filtration rate abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (2)
skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 3 (4)
hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
lipase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
malaise (General disorders) | 0 (0) | 0 (0) | 2 (2)
fatigue (General disorders) | 3 (3) | 4 (4) | 1 (1)
renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
peripheral neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
hallucination, visual (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (3)
abnormal weight gain (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
epigastric discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
urine bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
weight decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
hyper IgE syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
intrahepatic portal hepatic venous fistula (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT01968382/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT01968382/ICF_001.pdf